CLINICAL TRIAL: NCT04063137
Title: Black Rice Anthocyanin in Mixed Meals: Influence on Postprandial Glycaemic and Lipid Responses Among Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Mei Hui Liu, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/00971
Record Dates: First submitted 2019-06-20; First posted 2019-08-21 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2021-07

CONDITIONS: Postprandial Hyperglycemia; Lipidemia
Keywords: Black rice; Anthocyanin; Lipidemia; High-fat diet
MeSH Terms: conditions — Hyperglycemia; Hyperlipidemias | interventions — CD36 Antigens

STUDY DESIGN:
Intervention Model Description: This study is a within-subject cross-over trial design to assess the influence of black rice anthocyanin on postprandial blood glucose and insulinemic responses, and lipid profiles.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anthocyanin fortified bread (Active Comparator): White bread is fortified with a 25% (w/w) black rice anthocyanin extract. Extract fortification is 4% w/w of bread flour.
  Interventions: Dietary Supplement: Anthocyanin fortified bread with beef patty (35% fat)
- White bread (Placebo Comparator)
  Interventions: Dietary Supplement: Anthocyanin fortified bread with beef patty (35% fat)

INTERVENTIONS:
Dietary Supplement: Anthocyanin fortified bread with beef patty (35% fat) — Bread is fortified at a 4% level using 25% (w/w) anthocyanin black rice extract. It is served with a beef patty (35% fat) to simulate a high-fat diet.

SUMMARY:
The diabetes epidemic is a pertinent concern globally. The prevalence of this metabolic disease among adults had been disclosed by the World health Organisation (WHO), reporting a total of 422 million diabetic adults and 3.7 million diabetic deaths in 2016, with Asian countries contributing more than 60% of the world's diabetic population. Due to its economic and social repercussions, preventive strategies are implemented at a population level. The implementation of a diet low in glycaemic index (GI) has been widely adopted as part of diabetes management strategies to prevent and control Type 2 Diabetes Mellitus (T2DM) as the consumption of food with low GI has shown to improve glycaemic control, lipid profile, and reduce systemic inflammation. Other strategies include adopting an active lifestyle and the consumption of functional foods. In lieu of this, the composition of food products may be altered by incorporating edible plant-based functional components with carbohydrase-inhibiting properties. Black rice has been proposed as a viable source of functional ingredients, namely anthocyanins, not only because of its potential benefits to health that has been established by numerous in-vitro studies, but also it is easily sourced for in Asia as it is widely cultivated.

In this study, black rice anthocyanin-fortified bread serves as a replacement to white bread as the staple to the subject's diet, in a mixed meal setting. The fortified bread is hypothesised to improve glycemic responses over white bread, offering a lower GI food alternative to the conventional staple.

DETAILED DESCRIPTION:
Black rice anthocyanin-fortified bread, compared to white bread as a control, is hypothesised to improve glycaemic control and serum lipid profiles in a mixed meal setting. The aim of this research is to to assess the influence of black rice anthocyanin on postprandial blood glucose and insulinemic responses, and lipid profiles.

The aim of the research is to contribute to the prevention of diabetes by investigating how the incorporation of functional ingredients in carbohydrate-based foods will influence glycaemic and lipid panel profiles in a mixed meal setting. A human in-vivo intervention study will be conducted to assess the glycaemic and lipid responses of anthocyanin-fortified bread as compared to white bread, served with a ground beef patty to simulate the mixed meal. The approximate time to complete study recruitment will be 4 weeks.

Healthy, non-smoking subjects aged 21 to 65 will be recruited in this study. There will be a total of 2 visits (excluding 1 screening session), with the duration of each visit approximately 4-5 h. The study procedures will be conducted in Investigational Medicine Unit (IMU). During the each visit, subjects will undergo a mixed meal tolerance test. Test foods will be freshly prepared on the day of the visit in Food Science amp; Technology Programme food preparation area situated at Block S14 level 5, Science Drive 2, using food-grade ingredients. Only small quantities of bread will be prepared each day (3 to 4). The subject's glycemic response to the control meal (white bread) will be compared to their response after consumption of anthocyanin-fortified bread in a mixed meal setting. An improvement in postprandial blood glucose response and lipid panel profiles in response to the mixed meals will show that the anthocyanin-fortification is effective in offering better control over glycaemic and lipid profiles.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* Age between 21 - 65 years old.
* Healthy Body Mass Index (BMI) range of

  * males: >=18.5 kg/m2 and <=24.9 kg/m2,
  * females: >=18.5 kg/m2 and <=22.9 kg/m2.
* Overtly healthy males or females, as determined by medical history, physical examination and laboratory results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Males and females with stable medical problems that, in the investigator's opinion, will not significantly alter the performance of the biomarker panel, will not place the subject at increased risk by participating in the study, and will not interfere with interpretation of the data.
* Not on any regular medications (western/traditional medicine). Nutritional supplements with established chemical composition that can be ascertained and clearly recorded is acceptable. However, subjects using traditional medicine (with compositions that cannot be ascertained) will be excluded in this study.
* Have sufficient venous access to allow for blood sampling as per the protocol.
* Reliable and willing to make themselves available for the duration of the study, and are willing to follow study procedures.
* No dietary restriction to beef intake.

Exclusion Criteria:

* Persons with a history, or presence of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, malignancy or neurological disorders capable of significantly altering the performance of the biomarker panel; or of interfering with the interpretation of data.
* Persons with electronic medical implants (e.g. pacemaker).
* Persons with known or ongoing psychiatric disorders within 3 years.
* Persons with regular use of known drugs of abuse within 3 years.
* Women who are pregnant or lactating.
* Persons who have donated more than 500 mL of blood 4 weeks prior to study enrolment.
* Persons with an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females). 1 unit is equivalent to:

  * 12 oz or 360 mL of beer;
  * 5 oz or 150 mL of wine;
  * 1.5 oz or 45 mL of distilled spirits.
* Persons with uncontrolled hypertension (i.e. blood pressure >160/100 mmHg)
* Persons with active infection(s) requiring systemic, antiviral or antimicrobial therapy that will not be completed prior to the first study visit.
* Persons who have undergone treatment with any investigational drug or biological agent within one (1) month of screening, or plans to enrol in another study involving investigational drugs/ biological agents during the duration of this study.
* Persons with a known allergy to insulin.
* Persons with a history of bleeding diathesis or coagulopathy.
* Persons with fasting glucose of >=126 mg/dL (>=7 mmol/L) or 2-hour postprandial glucose of >=200 mg/dL (>=11.1 mol/L).
* Persons with clinically significant (as determined by investigator) abnormalities on laboratory examination that will increase risk to the subject or interfere with data integrity.
* Persons with any other conditions which, in the opinion of the Investigator, would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study.
* Persons with significant change in weight (+/- 5%) during the past month.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in area under curve for Low-density lipoprotein cholesterol (LDL-c) | 0 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 180 minutes, 240 minutes.
  mmol/L*min; area under curve

SECONDARY OUTCOMES:
Change in area under curve for Blood glucose | 0 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 180 minutes, 240 minutes.
  mmol/L*min; area under curve

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hui Liu, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Will be decided on a later date.